CLINICAL TRIAL: NCT01398540
Title: Characterisation of Cellular and Humoral Immunity in Elderly People After Immunization With a Purified, Inactivated Japanese Encephalitis Vaccine.
Brief Title: Cellular and Humoral Immunity in Elderly After Immunization With a Japanese Encephalitis Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Univ. Prof. Dr. Ursula Wiedermann, Univ.Prof. MD, PhD, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IX-sensesc 1.2
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Humoral and Cellular Immune Responses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- elderly (Experimental): subjects are at least 60 years old (with no upper age limit), receiving 2 immunisations with IXIARO
  Interventions: Biological: IXIARO
- young (Experimental): subjects 18 to 40 years old, receiving 2 immunisations with IXIARO
  Interventions: Biological: IXIARO

INTERVENTIONS:
Biological: IXIARO — 2 immunizations (0,5ml) with a 28 day interval

SUMMARY:
The aim of this project is to investigate humoral and cellular immune responses before and after immunisation with the Japanese encephalitis vaccine IXIARO in subjects above 60 years of age and 18-40 years old subjects.

ELIGIBILITY:
Inclusion Criteria:

* adults (18-40 years old)
* adults (≥60 years),
* both sexes
* willingness to sign written informed consent form

Exclusion Criteria:

* age below 18 years or between 41-59 years old
* status post japanese encephalitis, tick born encephalitis (TBE), dengue, yellow fever or West Nile virus infection
* previous immunization against yellow fever, japanese encephalitis (dengue or WNV)
* current acute infection (body temperature above 37,9°C)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
cellular immunity (cytokine production upon stimulation with Japanese Encephalitis (JE) Virus Antigen) 7 days after the 2. JE-vaccination | 7 days after the 2 JE vaccinations

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Wiedermann, MD, PhD, Principal Investigator — Institute of Specific Prophylaxis and Tropical medicine, Vienna